CLINICAL TRIAL: NCT00471172
Title: A 6-Month, Randomized Study To Evaluate The Efficacy Of Various Non-Pharmacologic, Disease Management Programs For The Treatment Of Obesity
Brief Title: Study of Five Different Methods Of Delivering A Lifestyle Modification Program for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A9001187
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Face-to-face counseling by a dietitian (months 1-3: weekly, months 4-6: every other week)
Behavioral: Face-to-face counseling by a dietitian (monthly)
Behavioral: Counseling by a dietitian via telephone (months 1-3: weekly, months 4-6: every other week)
Behavioral: Counseling by a dietitian via e-mail (months 1-3: weekly, months 4-6: every other week)
Behavioral: Self help

SUMMARY:
The aim of the study was to compare 5 methods of delivering a weight loss lifestyle modification program to obese patients on a background of sibutramine. The methods differed in the type and frequency of counseling utilized to deliver dietary, physical activity and behavioral recommendations for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 1- Body mass index -calculated as weight in kilograms divided by the square of height in meters- ≥30 and <40 kg/m2.
* 2- Eligibility to be prescribed sibutramine, following the eligibility requirements listed in the US Package Insert
* 3- Willingness and ability to comply with study related procedures
* 4- Access to Internet and email

Exclusion Criteria:

* Uncontrolled blood pressure (defined as ≥140/90 mmHg), diabetes, coronary heart disease, chronic congestive heart failure, stroke, significant metabolic, hepatic or renal disease, current malignancy, gastric bypass surgery or had a weight loss ≥10%, participated in a structured weight loss program, or had taken weight loss agents during the past 6 months. Women were excluded if pregnant or breastfeeding; women of childbearing potential had to use adequate contraception.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350
Dates: Start 2004-08; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight at 6 months.

SECONDARY OUTCOMES:
Changes in waist circumference, lipids, glucose, insulin, blood pressure, quality of life and weight-related symptoms at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Harleysville, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001187&StudyName=Study+of+Five+Different+Methods+Of+Delivering+A+Lifestyle+Modification+Program+for+Weight+Loss+